CLINICAL TRIAL: NCT03341390
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel Group Study to Evaluate the Effect of Coadministration of Multiple Doses of BMS-986177 on Aspirin in Healthy Participants
Brief Title: An Investigational Study to Assess the Effect of BMS-986177 on Aspirin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CV010-027
Record Dates: First submitted 2017-10-30; First posted 2017-11-14 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Healthy Volunteers
Keywords: Healthy participants; Healthy subjects; Strokes
MeSH Terms: conditions — Stroke | interventions — Aspirin; milvexian

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Aspirin (Active Comparator): 325 mg tablet, once daily for 5 days (Day -5 to -1)
  Interventions: Drug: Aspirin
- BMS-986177 plus aspirin (Experimental): 200 mg BMS-986177 twice daily and 325 mg tablet aspirin once daily (Day 1-7)
  Interventions: Drug: Aspirin; Drug: BMS-986177
- Placebo plus aspirin (Placebo Comparator): 200 mg Placebo twice daily and 325 mg tablet aspirin once daily (Day 1-7)
  Interventions: Drug: Aspirin; Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — 1 x 325 mg tablet of aspirin administered once daily
  Other Names: Acetylsalicylic Acid
Drug: BMS-986177 — 200 mg of BMS-986177 administered twice daily
  Arms: BMS-986177 plus aspirin
Drug: Placebo — 200 mg of Placebo administered twice daily
  Arms: Placebo plus aspirin

SUMMARY:
The purpose of this study is to investigate the effect of taking multiple doses of BMS-986177 when aspirin is taken once-daily. Eligible participants will receive twice-daily doses of BMS-986177 or placebo, with a once-daily dose of aspirin. The safety, tolerability and movement of BMS-986177 into, through and out of the body (pharmacokinetics/PK) will be assessed, as will the effect of BMS-986177 on the PK of aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent form.
* Healthy male and female participants (not of childbearing potential), determined by no clinically significant deviation from normal in medical history, physical examination, ECGs (electrocardiograms) and clinical laboratory determinations.
* Women participants must have documented proof they are not of childbearing potential.
* Males sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for duration of treatment with BMS-986177, and for a total of 93 days after the last dose of BMS-986177; and must be willing to refrain from sperm donation during this time. Azoospermic males are exempt from contraceptive requirements.
* Normal renal function at screening (Glomerula Filtration Rate ≥ 80 mL/min/1.73 m2.
* Body Mass Index (BMI) of 18.0 kg/m2 to 32.0 kg/m2 inclusive.

Exclusion Criteria:

* Women who are of childbearing potential or breastfeeding.
* Any significant acute or chronic illness.
* History of gastroesophageal reflux disease, dyspepsia, protracted nausea or chronic diarrhea.
* History of upper gastrointestinal ulcer disease within 6 months or current symptomatic or recent gastrointestinal disease that could impact absorption of study treatment.
* Abnormal renal profile and/or hematuria (if male) within 3 months of study start.
* History or evidence of abnormal bleeding and/or coagulation disorder and/or evidence of coagulopathy, prolonged or unexplained clinically significant bleeding, or frequent unexplained bruising or thrombus formation, or a history of spontaneous bleeding.
* Any major surgery within 4 weeks of study treatment administration or planned within 2 weeks after completion of the study.
* Donation of blood to a blood bank or in a clinical study (except screening or follow-up visit) within 4 weeks of study treatment administration (within 2 weeks for plasma only).
* Blood transfusion within 3 months of study treatment administration.
* Use of tobacco- or nicotine-containing products (including, but not limited to cigarettes, pipes, cigars, e-cigarettes, chewing tobacco, nicotine patches, nicotine lozenges or nicotine gum) within 6 months prior to study treatment administration.
* History of allergy to aspirin or related compounds.

Other protocol-defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs) leading to discontinuation when coadministered BMS-986177 (twice daily) and aspirin (once daily) | Up to 10 days
  Safety and tolerability of multiple doses of BMS-986177 measured by investigator assessment
Number of potential clinically significant changes in electrical activity of the heart in participants coadministered BMS-986177 (twice daily) and aspirin (once daily) | Up to 10 days
  Measured by electrocardiogram (ECG)
Number of participants with vital sign abnormalities. | Up to 10 days
Number of participants with physical examination abnormalities. | Up to 10 days
Number of participants with clinical laboratory abnormalities. | Up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Austin Clinic, Austin, Texas, United States

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx